CLINICAL TRIAL: NCT05026918
Title: A Comparison Between the Effectiveness of Manual Chest Physiotherapy and Active Cycle of Breathing Techniques (ACBT) in Patients of Cystic Fibrosis
Brief Title: Manual Chest Physiotherapy and Active Cycle of Breathing Techniques (ACBT) in Patients of Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/Lhr/0332 Hafsa Javed
Record Dates: First submitted 2021-08-27; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — S-(N-monomethoxytritylaminoethyl)-O-(2-chlorophenyl)phosphorothioate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): all the components of Manual Chest Physiotherapy wer performed on the patients of this group. MCPT was done few hours before meals and it was made sure that nothing was in patient's mouth while doing chest physiotherapy. MCPT includes postural drainage, percussion and vibrations. Chest Physiotherapy was done thrice a day for 30 minutes and there were 21 sessions a week.
  Interventions: Other: MCPT
- Group B (Experimental): all the components of Active Cycle of Breathing techniques (ACBT) were performed on the patients of this group. ACBT includes Breathing control techniques, chest expansion exercises and Forced Expiration Technique. These were performed thrice a day for 30 minutes and for 21 sessions a week.
  Interventions: Other: ACBT

INTERVENTIONS:
Other: MCPT — Postural Drainagewith percussion and vibration
  Arms: Group A
Other: ACBT — ACBT includes Breathing control techniques, chest expansion exercises and Forced Expiration Technique
  Arms: Group B

SUMMARY:
Cystic fibrosis is a genetic disease (autosomal recessive) which involves malfunction of the exocrine glands, leading to abnormal secretions in the body. It is a progressive disease that causes persistent lung infections and limits the ability to breathe over time. Clinical symptoms include persistent coughing, at times with phlegm, wheezing or shortness of breath, fatigue, difficulty with bowel movements sinus infections, poor growth, clubbing of the fingers and toes, and infertility in most males. The disease must be managed throughout life with diet, medication and preventive chest physical therapy as soon as any symptoms are noted in the young child. The purpose of the study was to evaluate the difference between the effects of Manual Chest Physiotherapy (CPT) and Active Cycle of Breathing Techniques (ACBT) in patients of Cystic Fibrosis. The tools of our study were Modified Borg Dyspnea Scale and Quality of well-being Scale. The total sample of our study was 14 out of which 7 were included in GROUP A and 7 Group B. SPSS 23 was used for statistical analysis and parametric tests were used for analysis

ELIGIBILITY:
Inclusion Criteria:

* Age limit 5-25
* Patients with confirmed diagnosis of Cystic Fibrosis
* Male and female.
* Clinically Stable Patients

Exclusion Criteria:

* Hypertensive patients.
* Intolerant patients.
* Compromised Renal Function.
* Other Comorbidities

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-07-04 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Modified Borg dyspnea Scale | 2nd week
  Modified Borg Dyspnea Scale is most commonly used to assess symptoms of breathlessness. It has a range from 0 to 10 (with 0 being no exertion and 10 being maximum effort).
Quality of well-being Scale | 2nd week
  The Quality of Well-Being Scale (QWB) is a general health quality of life questionnaire which measures overall status and well-being over the previous three days in four areas: physical activities, social activities, mobility, and symptom/problem complexes. It consists of 71 items and takes 20 minutes to complete

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- PAF Hospital, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalamara EI, Ballas ET, Pitsiou G, Petrova G. Pulmonary rehabilitation for cystic fibrosis: A narrative review of current literature. Monaldi Arch Chest Dis. 2021 Mar 11;91(2). doi: 10.4081/monaldi.2021.1501. PMID 33792230
- [Background] van der Schans C, Prasad A, Main E. Chest physiotherapy compared to no chest physiotherapy for cystic fibrosis. Cochrane Database Syst Rev. 2000;(2):CD001401. doi: 10.1002/14651858.CD001401. PMID 10796781
- [Background] Reisman JJ, Rivington-Law B, Corey M, Marcotte J, Wannamaker E, Harcourt D, Levison H. Role of conventional physiotherapy in cystic fibrosis. J Pediatr. 1988 Oct;113(4):632-6. doi: 10.1016/s0022-3476(88)80370-6. PMID 3171787
- [Background] Button BM, Wilson C, Dentice R, Cox NS, Middleton A, Tannenbaum E, Bishop J, Cobb R, Burton K, Wood M, Moran F, Black R, Bowen S, Day R, Depiazzi J, Doiron K, Doumit M, Dwyer T, Elliot A, Fuller L, Hall K, Hutchins M, Kerr M, Lee AL, Mans C, O'Connor L, Steward R, Potter A, Rasekaba T, Scoones R, Tarrant B, Ward N, West S, White D, Wilson L, Wood J, Holland AE. Physiotherapy for cystic fibrosis in Australia and New Zealand: A clinical practice guideline. Respirology. 2016 May;21(4):656-67. doi: 10.1111/resp.12764. Epub 2016 Apr 18. PMID 27086904
- [Background] McIlwaine MP, Lee Son NM, Richmond ML. Physiotherapy and cystic fibrosis: what is the evidence base? Curr Opin Pulm Med. 2014 Nov;20(6):613-7. doi: 10.1097/MCP.0000000000000110. PMID 25225791
- [Background] Bradley JM, Moran FM, Elborn JS. Evidence for physical therapies (airway clearance and physical training) in cystic fibrosis: an overview of five Cochrane systematic reviews. Respir Med. 2006 Feb;100(2):191-201. doi: 10.1016/j.rmed.2005.11.028. PMID 16412951
- [Background] Williams MT, Parsons DW, Frick RA, Ellis ER, Martin AJ, Giles SE, Grant ER. Acute respiratory infection in patients with cystic fibrosis with mild pulmonary impairment: comparison of two physiotherapy regimens. Aust J Physiother. 2001;47(4):227-36. doi: 10.1016/s0004-9514(14)60270-1. PMID 11722291
- [Background] Williams MT. Chest physiotherapy and cystic fibrosis. Why is the most effective form of treatment still unclear? Chest. 1994 Dec;106(6):1872-82. doi: 10.1378/chest.106.6.1872. No abstract available. PMID 7988215